CLINICAL TRIAL: NCT01004068
Title: Does Short-term Structured Exercise Training Program Plus Diet Intervention Improve Ovarian Sensitivity to Clomiphene Citrate in Polycystic Ovary Syndrome Patients (PCOS)? A Prospective Randomized Controlled Study
Brief Title: Short-term Structured Exercise Training Program Plus Diet Intervention in Patients With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Department of Obstetrics and Gynecology, University Magna Graecia of Catanzaro
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/2009
Record Dates: First submitted 2009-07-15; First posted 2009-10-29 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Polycystic Ovary Syndrome; Anovulation
Keywords: Clomiphene; Diet; Exercise; Infertility; PCOS; Physical activity; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Anovulation; Motor Activity; Infertility | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SET-diet plus clomiphene (Experimental): Structured exercise program plus hypocaloric diet for two months and received one-cycle of clomiphene citrate for one cycle
  Interventions: Other: SET-diet plus clomiphene
- Clomiphene citrate (Active Comparator): One month of observation followed by one-cycle of clomiphene citrate therapy
  Interventions: Drug: Clomiphene citrate
- SET plus diet (Experimental): Lifestyle modifications for two months.
  Interventions: Behavioral: Structured exercise program plus hypocaloric diet

INTERVENTIONS:
Other: SET-diet plus clomiphene — Two months of structured exercise program plus hypocaloric diet followed by 150 mg daily of clomiphene citrate
  Other Names: Lifestyle modification; CC
  Arms: SET-diet plus clomiphene
Drug: Clomiphene citrate — Clomiphene citrate at 150 mg daily for one cycle
  Other Names: CC
  Arms: Clomiphene citrate
Behavioral: Structured exercise program plus hypocaloric diet — SET plus diet
  Other Names: Lifestyle modifications
  Arms: SET plus diet

SUMMARY:
Clomiphene citrate (CC) is the first-line therapy for infertile women with polycystic ovary syndrome (PCOS). Unfortunately, at least 20% of PCOS results are not responsive to CC. Structured exercise training (SET) and diet has been successfully employed to restore ovarian function and to improve reproductive outcomes in obese and overweight women with PCOS. The current study was aimed to test the hypothesis that a short-term SET program plus diet intervention can improve the ovarian response to CC in CC-resistant PCOS patients.

DETAILED DESCRIPTION:
Ninety-six PCOS patients considered CC-resistant because not responsive to 150 mg daily of CC were randomized in three arms (group A, B, and C). Group A underwent SET program plus hypocaloric diet for two months, group B had one month of observation followed by one-cycle of CC therapy, and group C underwent SET program plus hypocaloric diet for two months and received one-cycle of CC for one cycle. CC was always given at the maximal dose previously used. Clinical, hormonal and metabolic data were assessed at baseline and after intervention. Ovulation was monitored by ultrasound and confirmed by plasma progesterone assay.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Anovulation

Exclusion Criteria:

* Major Medical Condition
* Severe Obesity

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Ovulation rate | three months

SECONDARY OUTCOMES:
Clinical data | three months
Metabolic data | three months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — University Magna Graecia
Locations (1):
- "Pugliese" Hospital, Catanzaro, Italy

REFERENCES:
- [Background] Vigorito C, Giallauria F, Palomba S, Cascella T, Manguso F, Lucci R, De Lorenzo A, Tafuri D, Lombardi G, Colao A, Orio F. Beneficial effects of a three-month structured exercise training program on cardiopulmonary functional capacity in young women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Apr;92(4):1379-84. doi: 10.1210/jc.2006-2794. Epub 2007 Jan 30. PMID 17264174
- [Background] Palomba S, Giallauria F, Falbo A, Russo T, Oppedisano R, Tolino A, Colao A, Vigorito C, Zullo F, Orio F. Structured exercise training programme versus hypocaloric hyperproteic diet in obese polycystic ovary syndrome patients with anovulatory infertility: a 24-week pilot study. Hum Reprod. 2008 Mar;23(3):642-50. doi: 10.1093/humrep/dem391. Epub 2007 Dec 23. PMID 18158291
- [Result] Palomba S, Falbo A, Giallauria F, Russo T, Rocca M, Tolino A, Zullo F, Orio F. Six weeks of structured exercise training and hypocaloric diet increases the probability of ovulation after clomiphene citrate in overweight and obese patients with polycystic ovary syndrome: a randomized controlled trial. Hum Reprod. 2010 Nov;25(11):2783-91. doi: 10.1093/humrep/deq254. Epub 2010 Sep 21. PMID 20858697